CLINICAL TRIAL: NCT04222036
Title: Turkish Validity and Reliability of the Expectation Scale in the Treatment of Chronic Pain
Brief Title: Validity and Reliability of the Expectation Scale in the Treatment of Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, aydan aytar, ASSOC. PROF., Baskent University
Other Study IDs: KA19/430
Record Dates: First submitted 2019-12-31; First posted 2020-01-09 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Musculoskeletal Disorder; Chronic Pain
Keywords: Reliability; Validity; Chronic Pain Treatment Expectations Scale; Turkish
MeSH Terms: conditions — Musculoskeletal Diseases; Chronic Pain | interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Translating the Questionnaire into Turkish and Related Processes — The first step is the translation from the original language to the other language. The ideal target in the translation phase is to use people who are familiar with the structure of the original language and who are familiar with the language. Two forward translation and one reverse translation methods will be applied after obtaining the written permission of the authors. After the completion of this phase, the terminological differences arising from the translators in the translation process from the original language to Turkish will be collected and discussed on the questions. The cultural adaptation study will be terminated by determining the equivalence between the Turkish version of the index and the English original. The final version of the questionnaire and the necessary changes will be arranged specific to the investigator's society and the authors of the original questionnaire will be consulted and the questionnaire will be finalized.
Other: Validity — The scale will be applied by face-to-face technique and convergent (moderate-high correlation with optimism measure) and distant (low correlation with depression and anxiety measures) validity will be evaluated.
Other: Reliability — The reliability of the materials will be tested with Cronbach alpha.

SUMMARY:
Questionnaires are available to measure expectations based on patient and treatment expectations in musculoskeletal disorders. In order to elucidate the factors that change expectations in the treatment of pain, more valid and reliable measurement tools are needed to measure the expectations of patients. The validity and reliability made in Turkey, there is no comprehensive study that measures the expectations of treatment. Therefore, the aim of this study was to test the Turkish validity and characteristics of the Chronic Pain Expectations Scale in patients with pain due to chronic musculoskeletal disorders.

DETAILED DESCRIPTION:
Considering the multidimensionality of pain experience, multidisciplinary approaches are accepted as gold standards in the treatment of pain . Pharmacological and non-pharmacological interventions, therapeutic therapies and treatment beliefs are generally considered to be key to these approaches. However, clinically significant pain treatment responses have not yet been clearly defined . Research suggests that their expectations may be one of the key components in the treatment of pain.

Expectation refers to the complex interplay of thoughts, values, and beliefs that are composed of past experiences and represent an assessment of expected outcomes specific to a situation. Four types of expectations have been proposed: ideal (desires and outcome preferences), predicted (expected outcome), normative (what one thinks should be) and unformed (not explicitly expressed). Numerous studies have demonstrated the importance of expectations in pain experience. Expecting pain reduction is usually associated with decreased pain intensity and improved treatment outcomes. In contrast, expecting increased pain is associated with increased pain. Complex and severe expectations may also affect treatment response. A person's level of participation in the treatment plan can be greatly influenced by expectations. Waiting for the full recovery of chronic pain as a result of treatment may pose an obstacle to functioning and quality of life.

Questionnaires are available to measure expectations based on patient and treatment expectations in musculoskeletal disorders. In order to elucidate the factors that change expectations in the treatment of pain, more valid and reliable measurement tools are needed to measure the expectations of patients. The validity and reliability made in Turkey, there is no comprehensive study that measures the expectations of treatment. Therefore, the aim of this study was to test the Turkish validity and characteristics of the Chronic Pain Expectations Scale in patients with pain due to chronic musculoskeletal disorders.

The study will be conducted on 198 volunteer individuals who apply to Baskent University Ankara Hospital Physical Medicine and Rehabilitation Department and will receive treatment due to chronic musculoskeletal diseases. Each individual participating in the study will be informed about the study.

Patients with pain due to chronic musculoskeletal disorders, native speakers of Turkish, those over the age of 18 and under 65 and literate individuals will be included in the study. Individuals with neurological disease and no pain problems will not be included in the study.

Treatment Expectations Scale in Chronic Pain, Positivity Scale, Hospital Anxiety and Depression Scale and Disease Cognition Questionnaire will apply.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pain due to chronic musculoskeletal disorders,
* native speakers of Turkish, those over the age of 18 and under 65 a

Exclusion Criteria:

* illiterate individuals
* Individuals with neurological disease and no pain problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who apply to Baskent University Ankara Hospital Physical Medicine and Rehabilitation Department and will receive treatment due to chronic musculoskeletal diseases.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-03-10 (Estimated)

PRIMARY OUTCOMES:
Treatment Expectations Scale in Chronic Pain | baseline
  The Chronic Pain Treatment Expectations Scale is a self-report questionnaire that measures the ideal and predicted expectations of patients. The items are designed to measure two aspects of expectations; ie process and result expectations. The instructions are as follows: The following questions are about your expectation for treatment for your chronic pain. For each question, please tick the box that is most appropriate, (1) What do you expect to be ideal during the healthcare appointment (s) (in the ideal world, what do you want it to happen) (2) What do you expect to be realistic during the healthcare appointment (s) (2) in real life, what do you actually expect). For each item, patients are asked to select the extent to which they will participate in an ideal and predicted expectations on a 5-point scale (1 = strongly disagree 5 = strongly agree). Thus, each item is scored twice by the participants.

SECONDARY OUTCOMES:
Positivity Scale | baseline
  Positivity Scale, directly evaluate the positivity levels of individuals. The original form of the instrument has a five-degree likert-type assessment. The Positivity Scale consists of eight items, one of which is reversed (item 6). internal consistency coefficient was found to be 0.75.
Hospital Anxiety and Depression Scale | baseline
  The aim of the scale is to determine the severity and severity of the patient by determining the patient's susceptibility to anxiety and depression. The test has a total of 14 questions. Seven of these questions measure anxiety (odd numbers) and the remaining seven measure depression (even numbers). The cut-off points were 10 for anxiety and 7 for depression. Accordingly, those above this score are considered at risk.
Disease Cognition Questionnaire | baseline
  Disease Cognition Questionnaire was determine the cognition of individuals. It is advantageous for large-scale operations due to its low cost, validity and reliability and ease of application. The questionnaire contains a list of statements of individuals with long-term illness. The questionnaire consists of 18 statements. Individuals are asked to what extent they accept the statements. 4 points indicate that they agree completely and 1 point indicates that they never agree. The expressions are grouped under 3 headings, 6 in each category;
  1. Helplessness (concentration on the deterrent aspects of the disease),
  2. Acceptance (a positive adaptation to chronic disease with emphasis on reducing its negative aspects),
  3. Perceived benefits (assigning positive meaning to the disease). High scores for the survey indicate that disease awareness is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided